CLINICAL TRIAL: NCT07230379
Title: Direct Visualization Endoscopic Retrograde Appendicitis Therapy (ERAT) Versus Laparoscopic Appendectomy (LA) for Acute Uncomplicated Appendicitis in Adults (E-APPEND): An Open-Label, Multicenter, Randomized Controlled Non-Inferiority Trial
Brief Title: Direct Visualization ERAT Versus Laparoscopic Appendectomy in Adults With Acute Uncomplicated Appendicitis
Acronym: E-APPEND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Micro-Tech (Nanjing) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhuan Liao, Zhuan Liao, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-APPEND
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Acute Uncomplicated Appendicitis
Keywords: ERAT; Endoscopic retrograde appendicitis therapy; Appendicitis; LA; Laparoscopic appendectomy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct Visualization ERAT (Experimental): Undergo direct visualization endoscopic retrograde appendicitis therapy
  Interventions: Procedure: Direct Visualization Endoscopic Retrograde Appendicitis Therapy
- Laparoscopic Appendectomy (Active Comparator): Undergo laparoscopic appendectomy
  Interventions: Procedure: Laparoscopic appendectomy

INTERVENTIONS:
Procedure: Direct Visualization Endoscopic Retrograde Appendicitis Therapy — Direct visualization ERAT will be performed by experienced endoscopists (≥ 30 prior ERAT cases) under conscious sedation or general anesthesia as needed. A colonoscope with a transparent cap will be advanced to the cecum to expose the appendiceal orifice, and a direct visualization appendicoscope will be introduced through the working channel. The appendiceal lumen will be inspected and irrigated with saline to clear pus and debris, with negative pressure applied for aspiration. Small appendicoliths will be flushed out, while larger ones will be removed using a retrieval basket, stone extractor, or laser lithotripsy. When narrowing or heavy purulence is present, a stent will be inserted for drainage. After confirming adequate drainage, the scope will be withdrawn. If ERAT fails, conversion to laparoscopic or open appendectomy will be performed.
  Other Names: ERAT
  Arms: Direct Visualization ERAT
Procedure: Laparoscopic appendectomy — Laparoscopic appendectomy will be performed under general anesthesia by surgeons with experience in > 20 procedures, according to standard clinical practice. The resected appendix will be examined for gross features and sent for histopathological confirmation of acute uncomplicated appendicitis. If laparoscopic appendectomy is unsuccessful, conversion to open appendectomy will be performed.
  Other Names: LA
  Arms: Laparoscopic Appendectomy

SUMMARY:
This study compares two ways of treating acute uncomplicated appendicitis, which is a mild form of appendicitis. In the Direct Visualization ERAT group, participants will receive Endoscopic Retrograde Appendicitis Therapy (ERAT). This is a minimally invasive, non-surgical treatment that uses a flexible endoscope passed through the colon to reach the appendix, clear the blockage, and drain the infection. In the Surgery group, participants will undergo Laparoscopic Appendectomy (LA), which is the current standard surgical treatment to remove the appendix. The purpose of this study is to determine whether ERAT is as safe and effective as standard surgery for treating uncomplicated appendicitis.

Before treatment, each participant will have a CT scan of the lower abdomen with contrast to confirm uncomplicated appendicitis and to rule out any signs of more serious infection. Participants will then be randomly assigned to either the ERAT group or the surgery group, and they will be informed of which treatment they will receive. Regardless of the group, all participants will receive the same supportive care, including pain relief, close monitoring, and a single dose of antibiotics before treatment. After the procedure, participants will stay in the hospital for at least 24 hours for observation. Follow-up will include an outpatient visit at 2 weeks, and telephone follow-ups at 1 month, 3 months, 6 months, and 1 year to monitor recovery and ensure that appendicitis does not recur.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized, non-inferiority trial comparing Direct Visualization Endoscopic Retrograde Appendicitis Therapy (ERAT) with Laparoscopic Appendectomy (LA) for the treatment of adult acute uncomplicated appendicitis (AUA). A total of 376 participants will be enrolled across 14 hospitals in China, and randomized in a 1:1 ratio to either ERAT or LA after providing informed consent.

Adults aged 18 years or older with CT-confirmed first-episode AUA are eligible. Key exclusions include complicated appendicitis, bowel obstruction, intolerance to colonoscopy or bowel preparation, poor operative candidacy, pregnancy, severe organ dysfunction, or concurrent participation in another clinical trial.

Interventions will be performed within 24 hours of admission. ERAT involves the use of a direct visualization appendicoscope to access the appendiceal lumen, irrigate pus and debris, and remove or fragment appendicoliths under direct vision. A short plastic stent may be placed if drainage is required. LA will be performed according to standard laparoscopic surgical techniques. Follow-up assessments will include an outpatient visit at 2 weeks and telephone follow-ups at 1, 3, 6, and 12 months.

The primary outcome is 30-day treatment success, defined as successful completion of the assigned procedure, resolution of symptoms, discharge without further surgery, and absence of recurrence. This study aims to provide robust evidence supporting the safety and effectiveness of ERAT and to inform future clinical guidelines for the management of acute uncomplicated appendicitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Diagnosis of first-episode acute uncomplicated appendicitis (AUA) confirmed by CT scan of the lower abdomen. AUA is defined as acute appendicitis without evidence of abscess, perforation, gangrene, or tumor.
3. Provision of written informed consent.

Exclusion Criteria:

1. Complicated appendicitis, defined as acute appendicitis with perforation, gangrene, periappendiceal abscess or phlegmon, generalized peritonitis, or radiologic evidence of extraluminal appendicolith, extraluminal air, periappendiceal fat stranding, or appendiceal mass.
2. Severe intestinal adhesions or bowel obstruction.
3. Intolerance or contraindication to bowel preparation or colonoscopy (e.g., intestinal perforation or bowel obstruction).
4. Poor general condition precluding tolerance of abdominal surgery.
5. Abdominal pain caused by other diseases as confirmed by CT or other diagnostic examinations, including inflammatory bowel disease, urinary tract disease, or gynecological disease.
6. Pregnancy.
7. Severe dysfunction of major organ systems, including but not limited to cardiac, pulmonary, renal, hepatic, or hematologic systems.
8. Current enrollment in another clinical trial.
9. Any condition that may prevent the participant from completing all study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Treatment Success | 30 days
  ERAT arm: Treatment success is defined as successful completion of the ERAT procedure, resolution of acute uncomplicated appendicitis symptoms, discharge from the hospital without appendectomy, and absence of recurrence within 30 days.
  LA arm: Treatment success is defined as successful completion of laparoscopic appendectomy without conversion to open appendectomy, histopathological confirmation of acute appendicitis characterized by the presence of neutrophilic infiltration within the appendiceal muscularis propria, resolution of acute uncomplicated appendicitis symptoms, and absence of recurrence within 30 days.

SECONDARY OUTCOMES:
Recurrence | 1 year
  Recurrent appendicitis defined as the occurrence of clinical symptoms consistent with appendicitis, leading to appendectomy after initial intervention, with histopathological confirmation of appendicitis in the resected appendix.
Technical success | Intraoperative
  ERAT arm: Successful endoscopic cannulation of the appendiceal orifice with appendicoscope insertion.
  LA arm: Completion of laparoscopic appendectomy without conversion to open surgery.
Timing to procedure | Pre-operative
  Measured in hours from the time of CT-confirmed diagnosis of AUA to the start of the procedure, as documented in the operative note.
Total procedure time | Intraoperative
  Represents the total time patient spent in the OR. Measured in minutes from the time the patient is wheeled into the operating room to the time the patient is wheeled out.
Intervention time | Intraoperative
  Measured in minutes from the beginning to the end of the intervention procedure, based on the operative note. For ERAT: from endoscope insertion to complete scope withdrawal. For LA: from skin incision to skin closure.
Preparation time | Intraoperative
  Defined as total procedure time minus intervention time. This duration includes time spent on equipment setup, administration of anesthesia, patient positioning, and draping.
Self-reported pain score | 1 month
  Assessed using the Visual Analogue Scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain).
Time to soft diet resumption | 1 week
  Number of days from the end of the procedure to patient-reported good tolerance of a soft diet. If soft diet is tolerated on the same day as the procedure, it will be recorded as 0 days.
Post-intervention narcotics used | 1 week
  Total amount of narcotics received during the primary hospitalization, both oral and intravenous, converted into intravenous morphine equivalents per kilogram of body weight.
Duration of analgesics used | 2 weeks
  Number of days from the end of the procedure to the last dose of analgesics (oral or intravenous) used for procedure-related abdominal pain.
Duration of post-intervention antibiotics used | 1 week
  Number of days from the end of the procedure to the last dose of prescribed antibiotics. Antibiotics may include both intravenous and oral forms. The day of the procedure is counted as Day 0.
Sick leave | 1 month
  Number of days participants are absent from work due to disease-related reasons, including post-intervention recovery.
Time to return to normal daily activities | 1 month
  The number of days it takes for participants to resume their normal everyday activities without significant discomfort after receiving the treatment.
Cost of treatment | 1 year
  Total direct hospital cost is calculated as the sum of all charges incurred, based on the hospital billing record.
Quality of Life of the Participants | 1 year
  Measured using the Chinese-validated EQ-5D-5L questionnaire.
Patient Satisfaction | 1 year
  Measured by the Global Assessment of Satisfaction, consisting of two questions:
  1. "How satisfied are you with the treatment you received for acute uncomplicated appendicitis?" Response on a 5-point Likert scale: very satisfied, satisfied, neutral, dissatisfied, very dissatisfied
  2. "Knowing how the treatment went, would you recommend it to someone else?" Response: Yes or No
Complication | 1 year
  Complications are defined as any adverse event related to the intervention (ERAT or LA). They will be classified as major or minor based on severity, according to the Clavien-Dindo classification system, with major complications defined as Clavien-Dindo Grade II or higher.

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Department of Gastroenterology, The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chingqing
  - Department of Gastrointestinal Surgery, The Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Department of Gastroenterology, South China Hospital, Medical School, Shenzhen University, Shenzhen, Guangdong
  - Department of Gastroenterology, The First Affiliated Hospital of Henan University,, Kaifeng, Henan
  - Department of Gastroenterology, The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Department of Gastrointestinal Surgery, Hunan Provincial People's Hospital, Changsha, Hunan
  - Department of Gastrointestinal Surgery, Xiangya Hospital, Central South University, Changsha, Hunan
  - Department of Gastrointestinal Surgery, The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Department of Gastroenterology, The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Department of Gastroenterology, Jilin City People's Hospital, Jilin, Jilin
  - Department of Gastroenterology, Linyi People's Hospital, Linyi, Shandong
  - Department of Gastrointestinal Surgery, Fourth West China Hospital, Sichuan University, Chengdu, Sichuan
  - Department of Gastrointestinal Surgery, The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Department of Gastroenterology, Changhai Hospital, Naval Medical University, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided
Undecided